CLINICAL TRIAL: NCT04245462
Title: Adequate Protein Intake Per Meal and Physical Disability in Mexican Adults Aged 60 Years and Older
Status: Completed | Type: Observational
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Collaborators: Hospital General de Occidente (Other)
Responsible Party: Principal Investigator, Juan Ricardo Lopez y Taylor, Director of the Institute of Applied Sciences for Physical Activity and Spor, Centro Universitario de Ciencias de la Salud, Mexico
Other Study IDs: HGO-ICAAFYD18-4
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Aging
Keywords: Protein intake; Older adults; Physical disability; Mexican adults

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Older aged (>60 years) Mexican adults attending to the Geriatrics Department from the Western General Hospital (Zapopan, Jalisco, Mexico).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Cross-sectional

SUMMARY:
This study sought to determine if the number of meals per day with an adequate protein content (defined as eating >30 g protein or >0.4 g protein/kg body mass each) is associated with presenting physical disability in Mexican adults aged 60 years and older. Physical disability was evaluated with self-reported questionnaires for different activities of daily living.

DETAILED DESCRIPTION:
Detailed dietary information was obtained for each participant to estimate dietary protein intake per meal (breakfast, lunch, dinner). One meal was considered with adequate protein content if it contained >30 g or >0.4 g/kg. Then, the number of meals with an adequate protein content was counted and classified as Zero meals, One meal, or Two or Three meals.

Physical disability was assessed with two validated questionnaires. One for instrumental activities of daily living (Lawton) and another for activities of daily living (Barthel). Disability was classified for each questionnaire item according to the authors' scales. Most items considered a physical disability if the participant reported any difficulty performing that task.

To analyze the association between the number of meals with adequate protein content (predictive variable) and physical disability (outcome variable), we used binomial logistic regression for each item. For the number of meals, we set the group of Zero meals as the reference. The analyses were adjusted for age, BMI categories, number of diagnosed diseases, sex, and inadequate protein intake per day (<1.2 g/kg/d).

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to stand up and walk independently or with walking sticks only.
* Subjects able to answer questionnaires independently or with minimum caregivers' assistance.

Exclusion Criteria:

* Subjects reporting any kind of hospitalization within the last year.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older aged Mexican adults attending to the Geriatrics Department at the Western General Hospital (Hospital General de Occidente) for their usual medical screening or first-time assessment.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Disability on Instrumental Activities of Daily Living | One day
  Disability reported for each item of instrumental activities of daily living (assessed with Lawton questionnaire). This instrument assesses how well the subject performs some daily activities involving tools (e.g. handling finances, taking medication, using the telephone). The instrument consists of five items for men and eight for women, and each item is coded for 0 (disabled) or 1 (functional) depending on if subjects are capable to successfully complete the activity. We only used the five items that apply for both men and women.

SECONDARY OUTCOMES:
Disability on Activities of Daily Living | One day
  Disability reported for each item of activities of daily living (assessed with Barthel questionnaire). This instrument assesses how well the subject performs some daily activities (e.g. dressing, using stairs). The instrument consists of ten items for both men and women coded as 0 or multiples of 5 (i.e. 5, 10, 15) depending on if subjects are capable to successfully complete the activity. When the subject performs the activity without difficulty (the highest score) he/she is deemed as functional, and any other difficulty as a disability.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gaytán-González, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Ciencias Aplicadas a la Actividad Física y al Deporte, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided